CLINICAL TRIAL: NCT05851742
Title: Effects of Myofascial Release With and Without Electrical Stimulation on Pain and Functionality in Women With Chronic Pelvic Pain
Brief Title: Effects of Myofascial Release and Electrical Stimulation in Chronic Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0507
Record Dates: First submitted 2023-03-31; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pelvic Pain; Myofascial Trigger Point Pain
Keywords: chronic pelvic pain syndrome; pelvic floor physical therapy; myofascial release; myofascial trigger points
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mfofascial release with electrical stimulation (Active Comparator): TENS 50-280 HZ frequency and a pulse duration of 50 us for 10 minutes along with 10 minutes myofascial release.
  Interventions: Device: TENS
- Myofascial release without electrical stimulation (Experimental): Release of trigger points
  Interventions: Other: Myofascial trigger point release

INTERVENTIONS:
Device: TENS — TENS 50-280 HZ frequency and a pulse duration of 50 us for 10 minutes along with 10 minutes myofascial release.
  Arms: Mfofascial release with electrical stimulation
Other: Myofascial trigger point release — Release of trigger points
  Arms: Myofascial release without electrical stimulation

SUMMARY:
Myofascial pelvic pain (MFPP) caused by myofascial trigger points (MTrPs) is a major contributor to chronic pelvic pain in women.In females,pelvic pain is the single most common indication for referral to women's health services.Pelvic floor physical therapy with myofascial release improve mobility and reduce pain by releasing the painful trigger points.Tools that will be used,for pain numerical pain scale (NPS),functional pelvic pain scale(FPPS) and pelvic floor impact questionnaire-7 will be used to asses pain and functionality.

DETAILED DESCRIPTION:
Myofascial pelvic pain (MFPP) caused by myofascial trigger points (MTrPs) is a major contributor to chronic pelvic pain in women. In females, pelvic pain ''is the single most common indication for referral to women's health services. Pelvic floor physical therapy with myofascial release improve mobility, and reduce pain by releasing the painful trigger points following restrictions in connective tissues that are related to pelvic floor.In this project we will observe effects of myofascial release with and without electrical stimulation on pain and functionality in women with chronic pelvic pain.It has been hypothesized that myofascial release along with electrical stimulation help in reducing pain and improve functionality in women.Patients will be having sessions for consecutive 4 weeks and will be exposed to both types of techniques to find out the effective results.

The study will be randomized control trial.For pain numerical pain scale (NPS),functional pelvic pain scale(FPPS) and pelvic floor impact questionnaire-7 will be used to asses pain and functionality respectively. A randomized control trial will be conducted on two groups. Group 1 will receive myofascial release with electrical stimulation in women with chronic pelvic pain for 4 weeks with 50-280 Hz frequency and a pulse duration of 50 µs for 10 minutes along with 10 minutes myofascial release..On the other hand Group 2 will receive myofascial release without electrical stimulation on pain and functionality in women with chronic pelvic pain. In previous studies there is ample amount of research conducted on chronic pelvic pain but there were very few recent studies available on myofascial release,so this relation of use of myofascial release with and without electrical stimulation on pain and functionality in chronic pelvic pain should also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-40 years,
* Presence of persistent chronic pelvic pain
* >4 points on a 10 point numeric rating scale for atleast more than 3 months,
* Atleast 1 active MTrp in one of the muscle groups including the obturator internus,
* levator ani,piriformis and coccygeus on pelvic examination.

Exclusion Criteria:

* Prolapse of the pelvic organ,
* Pregnency,
* Fibromyalgia

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
NPRS (Numeric Pain Rating Scale) | 4 weeks
  Higher the numeric value is 10 and lower is 0.The patient is asked to make three pain ratings corresponding to current,best and worst pain experienced over the past 24 hours on a scale of 0(no pain)to 10(worst pain imaginable).The average of the 3 ratings was used to represent the patient's level of pain over the previous 24 hours.
FPPS (Functional Pelvic Pain Scale) | 4 weeks
  Patients score pelvic function on the FPPS form for 8 categories:Bladder,Bowel,Intercourse,Walking,Running,Lifting,Working,Sleeping.The patients rated each category from 0 to 4,with 0 for normal function and 4 for cannot function because of pain.Thus each patient was given a total pelvic function score between 0 and 32.
PFIQ-7 (Pelvic Floor Impact Questionaire) | 4 weeks
  The PFIQ-7 consists of 7-questions that need to be answered 3 times each considering symptoms related to the Bladder or urine,Bowel or rectum,Vagina or pelvis and their effects on function,social health and mental health in the past 3 months.The responses for each question range from "Not at all-Somewhat-Moderately-Quit a bit". To get scale scores,the mean of each of the 3 scales is individually calculated,which ranges from 0 to 3,this number is then multiplied by 100 and then divided by 3.The scale scores are then added together to get the total PFIQ-7 score,which ranges from 0 to 300.A lower score means there is a lesser effect on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, MSWHPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shrikhande A, Ullger C, Seko K, Patil S, Natarajan J, Tailor Y, Thompson-Chudy C. A physiatrist's understanding and application of the current literature on chronic pelvic pain: a narrative review. Pain Rep. 2021 Aug 30;6(3):e949. doi: 10.1097/PR9.0000000000000949. eCollection 2021 Sep-Oct. PMID 34476302
- [Background] Castro-Sanchez AM, Gil-Martinez E, Fernandez-Sanchez M, Lara-Palomo IC, Nastasia I, de Los Angeles Querol-Zaldivar M, Aguilar-Ferrandiz ME. Manipulative therapy of sacral torsion versus myofascial release in patients clinically diagnosed posterior pelvic pain: a consort compliant randomized controlled trial. Spine J. 2021 Nov;21(11):1890-1899. doi: 10.1016/j.spinee.2021.05.002. Epub 2021 May 13. PMID 33991702
- [Background] Halder GE, Scott L, Wyman A, Mora N, Miladinovic B, Bassaly R, Hoyte L. Botox combined with myofascial release physical therapy as a treatment for myofascial pelvic pain. Investig Clin Urol. 2017 Mar;58(2):134-139. doi: 10.4111/icu.2017.58.2.134. Epub 2017 Feb 1. PMID 28261683
- [Background] Aredo JV, Heyrana KJ, Karp BI, Shah JP, Stratton P. Relating Chronic Pelvic Pain and Endometriosis to Signs of Sensitization and Myofascial Pain and Dysfunction. Semin Reprod Med. 2017 Jan;35(1):88-97. doi: 10.1055/s-0036-1597123. Epub 2017 Jan 3. PMID 28049214
- [Background] Fuentes-Marquez P, Cabrera-Martos I, Valenza MC. Physiotherapy interventions for patients with chronic pelvic pain: A systematic review of the literature. Physiother Theory Pract. 2019 Dec;35(12):1131-1138. doi: 10.1080/09593985.2018.1472687. Epub 2018 May 14. PMID 29757068
- [Background] Vural M. Pelvic pain rehabilitation. Turk J Phys Med Rehabil. 2018 Nov 4;64(4):291-299. doi: 10.5606/tftrd.2018.3616. eCollection 2018 Dec. PMID 31453525
- [Background] Sharma N, Rekha K, Srinivasan JK. Efficacy of transcutaneous electrical nerve stimulation in the treatment of chronic pelvic pain. J Midlife Health. 2017 Jan-Mar;8(1):36-39. doi: 10.4103/jmh.JMH_60_16. PMID 28458478
- [Background] Dal Farra F, Aquino A, Tarantino AG, Origo D. Effectiveness of Myofascial Manual Therapies in Chronic Pelvic Pain Syndrome: A Systematic Review and Meta-Analysis. Int Urogynecol J. 2022 Nov;33(11):2963-2976. doi: 10.1007/s00192-022-05173-x. Epub 2022 Apr 7. PMID 35389057
- [Background] Lewis GK, Chen AH, Craver EC, Crook JE, Carrubba AR. Trigger point injections followed by immediate myofascial release in the treatment of pelvic floor tension myalgia. Arch Gynecol Obstet. 2023 Apr;307(4):1027-1035. doi: 10.1007/s00404-022-06880-y. Epub 2022 Dec 14. PMID 36513896
- [Background] Natarajan J, Ahmed T, Patil S, Mamsaang M, Kapadia R, Tailor Y, Shrikhande A. Pain and functionality improved when underlying neuromuscular dysfunction addressed in chronic pelvic pain patients. Neurourol Urodyn. 2021 Aug;40(6):1609-1615. doi: 10.1002/nau.24726. Epub 2021 Jun 3. PMID 34082473
- [Background] Ajimsha MS, Ismail LA, Al-Mudahka N, Majzoub A. Effectiveness of external myofascial mobilisation in the management of male chronic pelvic pain of muscle spastic type: A retrospective study. Arab J Urol. 2021 Jul 26;19(3):394-400. doi: 10.1080/2090598X.2021.1954414. eCollection 2021. PMID 34552791
- [Background] Cottrell AM, Schneider MP, Goonewardene S, Yuan Y, Baranowski AP, Engeler DS, Borovicka J, Dinis-Oliveira P, Elneil S, Hughes J, Messelink BJ, de C Williams AC. Benefits and Harms of Electrical Neuromodulation for Chronic Pelvic Pain: A Systematic Review. Eur Urol Focus. 2020 May 15;6(3):559-571. doi: 10.1016/j.euf.2019.09.011. Epub 2019 Oct 19. PMID 31636030
- [Background] Mahran A, Baaklini G, Hassani D, Abolella HA, Safwat AS, Neudecker M, Hijaz AK, Mahajan ST, Siegel SW, El-Nashar SA. Sacral neuromodulation treating chronic pelvic pain: a meta-analysis and systematic review of the literature. Int Urogynecol J. 2019 Jul;30(7):1023-1035. doi: 10.1007/s00192-019-03898-w. Epub 2019 Mar 14. PMID 30874835
- [Background] Grinberg K, Weissman-Fogel I, Lowenstein L, Abramov L, Granot M. How Does Myofascial Physical Therapy Attenuate Pain in Chronic Pelvic Pain Syndrome? Pain Res Manag. 2019 Dec 12;2019:6091257. doi: 10.1155/2019/6091257. eCollection 2019. PMID 31915499
- [Background] Tam J, Loeb C, Grajower D, Kim J, Weissbart S. Neuromodulation for Chronic Pelvic Pain. Curr Urol Rep. 2018 Mar 26;19(5):32. doi: 10.1007/s11934-018-0783-2. PMID 29582185
- [Background] Baltazar MCDV, Russo JAO, De Lucca V, Mitidieri AMS, da Silva APM, Gurian MBF, Poli-Neto OB, Rosa-E-Silva JC. Therapeutic ultrasound versus injection of local anesthetic in the treatment of women with chronic pelvic pain secondary to abdominal myofascial syndrome: a randomized clinical trial. BMC Womens Health. 2022 Aug 2;22(1):325. doi: 10.1186/s12905-022-01910-y. PMID 35918696
- [Background] Modarresi S, Lukacs MJ, Ghodrati M, Salim S, MacDermid JC, Walton DM; CATWAD Consortium Group. A Systematic Review and Synthesis of Psychometric Properties of the Numeric Pain Rating Scale and the Visual Analog Scale for Use in People With Neck Pain. Clin J Pain. 2021 Oct 26;38(2):132-148. doi: 10.1097/AJP.0000000000000999. PMID 34699406
- [Background] Plavnik K, Tenaglia A, Hill C, Ahmed T, Shrikhande A. A Novel, Non-opioid Treatment for Chronic Pelvic Pain in Women with Previously Treated Endometriosis Utilizing Pelvic-Floor Musculature Trigger-Point Injections and Peripheral Nerve Hydrodissection. PM R. 2020 Jul;12(7):655-662. doi: 10.1002/pmrj.12258. Epub 2019 Nov 15. PMID 31587480